CLINICAL TRIAL: NCT01820078
Title: Effect of Paricalcitol on Albuminuria, Inflammation and Fibrosis on Proteinuric Chronic Renal Diseases (PALIFE Study): a Randomized Study
Brief Title: Paricalcitol on Albuminuria, Inflammation and Fibrosis on Proteinuric Chronic Renal Diseases (PALIFE Study)
Acronym: PALIFE
Status: Terminated | Phase: Phase 4 | Type: Interventional
Why Stopped: Recruitment not reached
Sponsor: Fundación Renal Iñigo Alvarez De Toledo (Other)
Collaborators: Effice Servicios Para la Investigacion S.L. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: PALIFE-2011-01
Record Dates: First submitted 2012-07-30; First posted 2013-03-28 (Estimated); Last update posted 2013-11-28 (Estimated); Status verified 2013-11

CONDITIONS: Chronic Kidney Disease, Unspecified
Keywords: Chronic; Kidney; Disease; Proteinuria; Albuminuria; Paricalcitol
MeSH Terms: conditions — Renal Insufficiency, Chronic; Bronchiolitis Obliterans Syndrome; Disease; Proteinuria; Albuminuria | interventions — Therapeutics

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Paricalcitol, Daily treatment, CKD (Experimental): Experimental Arm
  Interventions: Drug: Experimental arm; Other: Comparator Arm
- Daily treatment for CKD (Other): Comparator Arm
  Interventions: Other: Comparator Arm

INTERVENTIONS:
Drug: Experimental arm — Oral paricalcitol, 1 ug/day, plus daily treatment. 6 months (all study)
  Other Names: Treatment
  Arms: Paricalcitol, Daily treatment, CKD
Other: Comparator Arm — Daily treatment is not define by protocol, because daily treatment in CKD is highly variable and includes salt and/or blood pressure regulation, angiotensine system stoppers, controlled diet, etc.
  Other Names: Daily treatment for CKD

SUMMARY:
The purpose of this study is to estimate the differences between albuminuria values determined as Urine Albumin-to-Creatinine Ratio (UACR)(log transformed) from baseline to last observation caused by paricalcitol between the group of control and group of treatment.

DETAILED DESCRIPTION:
Clinical Trial to estimate UACR determined albuminuria differences between treatment and non-treatment groups from basal intake to last study-related observation. Patients should suffer proteinuric Chronical Kidney Disease and recovered levels of seric 25(OH)D. Also, this clinical trial tries to determinate the effect of paricalcitol over several metabolic and inflammatory parameters on patients.

ELIGIBILITY:
Inclusion Criteria:

* Informed consent signed
* Patients will be men or women, between 18 and 75 years old.
* Patients must have been taken an stable dosis of Angiotensine Converter Enzyme Inhibitor, Angiotensine Receptor Antagonism or antialdosterone at last 6 months before screening visit.
* Patients should not be on dialysis treatment.
* Women should not be pregnant, or in fertile period (at last 1 year postmenopausal or chirurgic sterilized or using this contraceptive methods: condoms, gel, intrauterine devices, anticonceptives, etc. During at last 3 months after the study beginning.

Exclusion Criteria:

* Patients have taken active vitamin D during 6 months after the screening.
* Patients with allergy o sensibility to paricalcitol.
* Patients with acute CKD 12 weeks before the screening.
* Patients with chronical gastrointestinal disease.
* Patients with hypo or hyperthyroidism.
* Patients with secondary hypertension
* Bad controled hypertension patients
* Patients with renal lithiasis
* Patients with drug dependence
* Patients taking calcitonins, biphosphonates, cinacalcet or others Ca-metabolism drugs.
* Patients taking immunosuppressor drugs.
* Patients not adequate to study as medical opinion.
* HIV patients
* Seric P > 5.0 mg/dl.
* Seric Ca> 10,0 mg/dl.
* Proteinuria > 3.500 mg/g
* Hypoalbuminemia < 3g/dl

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 127 (Actual)
Dates: Start 2012-05; Primary Completion 2013-09 (Actual); Study Completion 2013-12 (Estimated)

PRIMARY OUTCOMES:
Albuminuria in proteinuric Chronical Kidney Disease patients | 1 year
  Estimate differences between groups based on albuminuric level determined as UACR from basal to last observation visit.

SECONDARY OUTCOMES:
Change from baseline albuminuria at 6 months | 6 months
  Determinate % of patients with an over 20% of albuminuria descent from baseline

CONTACTS AND LOCATIONS:
Overall Officials: Jesús Egido de los Ríos, MD, Principal Investigator — Fundación Renal Iñigo Alvarez De Toledo
Locations (25):
- Spain (25):
  - Hospital Universitario General de Alicante, Alicante, Alicante
  - Hospital Son Espases, Mallorca, Balearic Islands
  - Hospital Germans Trias i Pujol, Badalona, Barcelona
  - Fundació Puigvert, Barcelona, Barcelona
  - Hospital Valle de Hebrón, Barcelona, Barcelona
  - Hospital de Galdakao, Bilbao, Basque Country
  - Hospital Virgen de la Candelaria, Santa Cruz de Tenerife, Canary Islands
  - Hospital Reina Sofía, Córdoba, Córdoba
  - Hospital Virgen de las Nieves, Granada, Granada
  - Hospital Comarcal Da Costa, Burela de Cabo, Lugo
  - Hosp. U. Fundación de Alcorcón, Alcorcón, Madrid
  - Hospital Gregorio Marañon, Madrid, Madrid
  - Hospital Ramon y Cajal, Madrid, Madrid
  - Clínico San Carlos, Madrid, Madrid
  - Fundación Jiménez Díaz, Madrid, Madrid
  - Hospital 12 de Octubre, Madrid, Madrid
  - Hospital Universitario La Paz, Madrid, Madrid
  - Hospital Universitario Puerta de Hierro, Majadahonda, Madrid
  - Hospital Infanta Sofía, San Sebastián de los Reyes, Madrid
  - Hospital Carlos Haya, Málaga, Málaga
  - Hospital Universitario Virgen de la Macarena, Seville, Sevilla
  - Hospital Universitario Virgen del Rocío, Seville, Sevilla
  - Hospital General Universitario de Valencia, Valencia, Valencia
  - Hospital Dr Peset, Valencia, Valencia
  - Hospital Clinico Lozano Blesa, Zaragoza, Zaragoza